CLINICAL TRIAL: NCT07222280
Title: Clinical Trial Protocol: Alzheimer's Dementia Underlying Encephalopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Covenant Health, US (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ADUE2025
Record Dates: First submitted 2025-07-21; First posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer Dementia; Alzheimer Disease; Delirium Confusional State; Encephalopathy; Cognitive Abnormality
MeSH Terms: conditions — Alzheimer Disease; Confusion; Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All eligible patients will receive a Quest AD-Detect blood test (Other): All patients that meet the inclusion criteria, and none of the exclusion criteria, will have their blood tested with the Quest AD-Detect
  Interventions: Diagnostic Test: Quest AD-Detect blood test

INTERVENTIONS:
Diagnostic Test: Quest AD-Detect blood test — Blood will be collected and sent for testing using the Quest AD-Detect blood test

SUMMARY:
The goal of this clinical trial is to determine if utilizing the Quest AD-Detect blood test, while patient's are hospitalized for a cognitive diagnosis (such as delirium or encephalopathy), will result in an earlier diagnosis of underlying Alzheimer's disease.

* Will this blood test have the ability to distinguish between Alzheimer's disease and other causes of cognitive impairment in the inpatient setting?
* Neurology Clinic will complete a 6-month post-hospitalization follow up with patients who have had the Quest AD-Detect Alzheimer's Disease blood test completed while they were inpatient to discuss the risk assessment portfolio

ELIGIBILITY:
Inclusion Criteria:

* Ages 60 to 90 years old
* No prior diagnosis of dementia
* Currently hospitalized with cognitive diagnosis, including but no limited to; delirium, encephalopathy, etc. thought to be secondary to a toxic/metabolic state

Exclusion Criteria:

* Age under 60 years
* Prior diagnosis of dementing illness or other organic etiology to cognitive impairment

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
To show the percentage of patients (21 patients in the study) who presented with a cognitive diagnosis (including but not limited to delirium, encephalopathy, etc.) that have a positive biomarker for Alzheimer's dementia | From enrollment to 6 month follow up appointment with Neurology Clinic.
  A Six month follow up with the Neurology clinic to discuss the results of Quest AD Detect (p-tau217), those patients who are found to have a positive outcome will receive additional follow-up in the Neurology clinic (which could include the use of additional lab tests or further diagnostic testing).

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Moore, MD, Principal Investigator — Covenant Health, Canada
Locations (6):
- United States (6):
  - Cumberland Medical Center, Crossville, Tennessee
  - Roane Medical Center, Harriman, Tennessee
  - Fort Sanders Regional Medical Center, Knoxville, Tennessee
  - Fort Loudon Medical Center, Lenoir City, Tennessee
  - Methodist Medical Center, Oak Ridge, Tennessee
  - LeConte Medical Center, Sevierville, Tennessee

IPD SHARING:
Plan to Share IPD: No